CLINICAL TRIAL: NCT05789758
Title: Spinraza (Nusinersen) SMA Pregnancy Exposure Study Within Existing SMA Registries
Brief Title: A Study to Learn How Nusinersen (Spinraza) Affects Participants With Spinal Muscular Atrophy (SMA) Who Took it Before or During Pregnancy And About The Health of Their Babies
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CH-SPN-12180; 232SM405 (Other: Biogen)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nusinersen Treated Participants: Pregnant participants with SMA who are exposed to nusinersen during the relevant window defined as 14 months prior to the first day of the participant's last menstrual period before conception, 14.5 months before conception and anytime during pregnancy and are enrolled in the registries, International Spinal Muscular Atrophy Registry (ISMAR), Adult SMA REACH and SMArtCARE will be followed prospectively up to 3 months post-delivery, the infants will be followed up to 2 years post-delivery and the available data is collected retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Administered as specified in the treatment arm.

SUMMARY:
In this study, researchers will know more about the effects of nusinersen, also known as Spinraza®, in pregnant participants with spinal muscular atrophy, also known as SMA. This is a drug available for doctors to prescribe for people with SMA. Due to the current treatment options that exist, people with SMA may now reach the age where they can become pregnant. But, there is not enough information known yet about what the effects of nusinersen may be on pregnant people with SMA or on their babies.

This is known as an "observational" study, which collects health information about study participants without changing their medical care. The pregnant participants for this study will be found using 3 different groups of SMA study research centers:

* ISMAR-US (International SMA Registry in the United States)
* UK Adult SMA-REACH (Adult SMA Research and Clinical Hub in the United Kingdom)
* SMArtCARE (Austria, Germany, and Switzerland)

The main goal of this study is to collect birth and health information from 3 groups of participants and their babies. These groups are:

* Those who received nusinersen 14 months before the first day of their last period before getting pregnant
* Those who received nusinersen 14.5 months before the day they got pregnant
* Those who received nusinersen during any time in their pregnancy

The main questions researchers want to learn about in this study are:

* Loss of pregnancy overall
* Loss of pregnancy before the baby was 20 weeks old
* Loss of pregnancy after the baby becomes 20 weeks old
* Live births
* Loss of the baby after birth
* Babies who have problems in their body that develop during pregnancy
* Babies who are small for their age while in the participant's uterus
* Pregnancy that happens outside of the uterus
* How many participants die during pregnancy, while the baby is being born, and up to 12 weeks after delivering the baby
* Babies who develop problems in their body after birth

Researchers will also compare this information to people without SMA who have not received nusinersen.

This study will be done as follows:

* Information will start being collected when the participant decides to join the study.
* Participants will be contacted at each trimester (about every 3 months) to learn about their health and pregnancy.
* Participants' doctors will be contacted at each trimester, when the participants are about 6 or 7 months pregnant, and about 4 weeks after the delivery of the baby.
* The babies' doctors will be contacted when the baby is 1, 2, 6, 12, 18, and 24 months old.
* Each participant will be in the study until the end of their pregnancy and for up to 12 weeks after delivery. Each baby will be in the study for up to 2 years after birth.
* The study overall will last at least 10 years from when the first participant joins the study.

DETAILED DESCRIPTION:
The primary objectives of the study are to prospectively evaluate pregnancy complications and outcomes in participants with SMA, birth outcomes and adverse effects in infants born to participants with SMA, who were exposed to nusinersen up to 14 months prior to the first day of their last menstrual period (LMP) before conception, 14.5 months before the date of conception, and/or at any time during their pregnancy. The secondary objective of the study is to evaluate pregnancy outcomes in participants with SMA exposed to nusinersen as compared with participants without SMA who were not exposed to nusinersen (e.g., participants from external, general population comparators).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant who is currently pregnant (or was pregnant during the relevant exposure window) and enrolled in the United States (US) network of the ISMAR registry, the United Kingdom (UK) Adult SMA REACH, or the Germany, Austria, or Switzerland network of the SMArtCARE registry
* Genetic documentation of spinal muscular atrophy linked to chromosome 5q (5q SMA)
* Documentation that the participant was exposed to nusinersen up to 14 months prior to the first day of their LMP before conception, 14.5 months before conception, and/or at any time during their pregnancy

Key Exclusion Criteria:

* Treatment with risdiplam at any time from the first day of their LMP, 2 weeks prior to the date of conception (approximately 5 half-lives), and/or plans to receive treatment with risdiplam during pregnancy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant participants with SMA who are exposed to nusinersen from the UK Adult SMA REACH, ISMAR - US, and SMArtCARE registries will be enrolled to obtain information on effects of nusinersen on pregnancy complications and outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Pregnancy Terminations | Up to 10 years
  Pregnancy termination is defined as any induced or voluntary fetal loss during pregnancy.
Number of Spontaneous Abortions | Up to 10 years
  Spontaneous abortion is defined as any loss of a fetus due to natural causes at <20 weeks of gestation.
Number of Fetal Deaths | Up to 10 years
  Fetal deaths include early fetal loss which is fetal death occurring at ≥20 weeks but <28 weeks of gestation and late fetal loss which is fetal death occurring at ≥28 weeks of gestation.
Number of Live Births | Up to 10 years
  Live births include premature births which is defined as delivery at <37 weeks of gestation, full term birth which is defined as delivery at ≥37 weeks of gestation.
Number of Neonatal, Perinatal, and Infant Deaths | Up to 10 years
  Neonatal death is defined as death occurring in a newborn prior to 28 days after birth. Perinatal death is defined as death occurring at or after 28 days and prior to 12 weeks after birth. Infant death is defined as death occurring between 12 and 52 weeks after birth, inclusive.
Number of Major Congenital Malformations (MCMs) | Up to 10 years
  MCMs (interchangeably referred to as congenital malformations, congenital anomalies, and birth defects) are abnormalities in structural development that are medically or cosmetically significant, are present at birth, and persist in postnatal life unless or until repaired.
Number of Infants Small for Gestational Age Birth | Up to 10 years
  Birth weight will be classified as small for gestational age (<10th percentile), appropriate (10th-90th percentile), or large (>90th percentile).
Number of Ectopic and Molar Pregnancies | Up to 10 years
  Ectopic pregnancy is defined as a pregnancy that occurs outside of the uterine cavity. Molar pregnancy is defined as genetically abnormal conceptions characterized by abnormal chorionic villi, trophoblastic hyperplasia, poor fetal development, and an increased risk of malignant disease development.
Number of Maternal Deaths | Up to 10 years
  Maternal deaths during pregnancy, labor, delivery, or up to 12 weeks after delivery will be reported.
Number of Infants With Abnormal Postnatal Growth and Development and Neurobehavioral Impairment | Up to 10 years
  Abnormal postnatal growth and development and neurobehavioral impairment in infants up to 24 months of age will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (2):
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Research Site, Cambridge, Massachusetts
- United Kingdom (9):
  - St George's University NHS Foundation Trust, London, Greater London
  - The Northern Care Alliance NHS Foundation Trust, Salford, Greater Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Nottingham University Hospitals Trust, Nottingham, Nottinghamshire
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - North Bristol NHS Trust, Bristol

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/